CLINICAL TRIAL: NCT06226415
Title: A Randomized Controlled Trial For Exploration of Stellate Ganglion Block in Patients With Cerebral Small Vessel Disease
Brief Title: Exploration of Stellate Ganglion Block in Patients With Cerebral Small Vessel Disease
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Zeng Changhao (Other)
Responsible Party: Sponsor-Investigator, Zeng Changhao, Research Director, People's Hospital of Zhengzhou University
Organization: People's Hospital of Zhengzhou University (Other)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 2024-KY-0118
Record Dates: First submitted 2024-01-18; First posted 2024-01-26 (Actual); Last update posted 2024-06-12 (Actual); Status verified 2024-06

CONDITIONS: Cerebral Small Vessel Diseases
MeSH Terms: conditions — Cerebral Small Vessel Diseases | interventions — Rehabilitation; Lidocaine

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- The comparison group (Active Comparator): The study lasted 14d for each patient. During the treatment, All the participants were provided with the rehabilitation therapy, which included routine rehabilitation, cognitive training, swallowing function training and nutrition support.
  Interventions: Behavioral: Rehabilitation therapy
- The observation group (Experimental): The study lasted 14d for each patient. During the treatment, All the participants were provided with the rehabilitation therapy, which included routine rehabilitation, cognitive training, swallowing function training and nutrition support.
  Based on the invention above, the patients in the observation group were provided, using 1.5ml of 2% Lidocaine hydrochloride (1ml: 0.5mg) and 500ug of Vitamin B12 (1ml: 0.5g).
  Interventions: Behavioral: Rehabilitation therapy; Procedure: Stellate ganglion block; Drug: Lidocaine Hydrochloride

INTERVENTIONS:
Behavioral: Rehabilitation therapy — The study lasted 14d for each patient. During the treatment, All the participants were provided with the rehabilitation therapy, which included routine rehabilitation, cognitive training, swallowing function training and nutrition support.
  Particularly, due to dysphagia, the patients enrolled might face difficulty in eating. For patients who were able to finish intake via mouth by compensatory means, the consistency, type, and size of food bolus was arranged. For those who cannot acquire sufficient nutrition through oral intake, the nasogastric tube feeding was provided.
Procedure: Stellate ganglion block — Based on the invention above, the patients in the observation group were provided with Stellate ganglion block, using 1.5ml of 2% Lidocaine hydrochloride (1ml: 0.5mg) and 500ug of Vitamin B12 (1ml: 0.5g). The percutaneous approach via the paratracheal route was used for Stellate ganglion block. The operator stood on the side of the block, instructed the patient to lie supine with a thin pillow placed below the shoulders, and tilted the head 45° towards the blocked side, fully exposing the neck. Then, routine disinfection of the neck skin was performed. The puncture site was located 2.5 cm above the sternoclavicular joint and 1.5 cm lateral to the midline of the neck.
  Arms: The observation group
Drug: Lidocaine Hydrochloride — Based on the invention above, the patients in the observation group were provided with Stellate ganglion block, using 1.5ml of 2% Lidocaine hydrochloride (1ml: 0.5mg) and 500ug of Vitamin B12 (1ml: 0.5g). The percutaneous approach via the paratracheal route was used for Stellate ganglion block. The operator stood on the side of the block, instructed the patient to lie supine with a thin pillow placed below the shoulders, and tilted the head 45° towards the blocked side, fully exposing the neck. Then, routine disinfection of the neck skin was performed. The puncture site was located 2.5 cm above the sternoclavicular joint and 1.5 cm lateral to the midline of the neck.
  Other Names: Lidocaine
  Arms: The observation group

SUMMARY:
This is a prospective study conducted on patients with Cerebral Small Vessel Disease, dysphagia and cognitive impairment. They were divided into the comparison group and observation group evenly. All the patients were provided with routine therapy, while the patients in the observation group were given Stellate Ganglion Block. The swallowing function, cognitive function and activities of daily living of the two groups of patients before and after treatment were evaluated by Penetration-Aspiration Scale, Mini-mental state examination and modified Barthel index.

DETAILED DESCRIPTION:
This study is conducted for Exploration of Stellate Ganglion Block in Patients With Cerebral Small Vessel Disease. This is a prospective study conducted on patients with Cerebral Small Vessel Disease, dysphagia and cognitive impairment. They were divided into the comparison group and observation group evenly. All the patients were provided with routine therapy, while the patients in the observation group were given Stellate Ganglion Block. The swallowing function, cognitive function and activities of daily living of the two groups of patients before and after treatment were evaluated by Penetration-Aspiration Scale, Mini-mental state examination and modified Barthel index.

ELIGIBILITY:
Inclusion Criteria:

* Age>18 years.
* Meeting the diagnostic criteria for cerebral small vessel disease.
* Dysphagia confirmed by Videofluoroscopic Swallowing Study
* Mini-Mental State Examination (MMSE)<27, indicating the existence of cognitive impairment.
* No history of prior stroke.
* Stable vital signs.

Exclusion Criteria:

* Dysphagia that might be caused by other diseases that might cause dysphagia, such as head and neck tumors, traumatic brain injury, myasthenia gravis, etc.
* Cognitive impairment that might be caused by other diseases, such as Alzheimer's disease, Parkinson's disease, brain injury, etc.
* Neurological blockade contraindications such as bleeding tendency, blocked site infection.
* Unable to successfully finish the assessment of this study.
* Complicated with severe liver and kidney failure, tumors, or hematological disorders.
* Simultaneously in need to undergo other therapy that might affect the outcomes of this study.
* Pregnant or nursing females

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 84 (Actual)
Dates: Start 2024-01-20 (Actual); Primary Completion 2024-05-25 (Actual); Study Completion 2024-06-01 (Actual)

PRIMARY OUTCOMES:
Penetration-Aspiration Scale | day 1 and day 14
  On the day 1 and day 14, Penetration-Aspiration Scale was used to assess dysphagia under Videofluoroscopic Swallowing Study, primarily evaluating the extent to which fluid food entered the airway and caused penetration or aspiration during the swallowing process. As the level increased, the severity of dysphagia also increased.

SECONDARY OUTCOMES:
Modified Barthel Index | day 1 and day 14
  On the day 1 and day 14, the activities of daily living of patients were assessed using the modified Barthel Index . The scale included 10 items such as feeding, bathing, walking, dressing. Each item was rated on a 4-point scale based on the level of assistance required, with a total score of 100 points. There was a positive correlation between activities of daily living and the final score.
Mini-Mental State Examination | day 1 and day 14
  On the day 1 and day 14, the cognitive function of patients was assessed using the Mini-Mental State Examination (MMSE). The MMSE evaluated five aspects, including orientation, memory, attention and calculation abilities, recall ability, and language skills, with a total score of 30 points. A MMSE score of less than 27 indicated cognitive impairment, with scores ≤9 indicating severe impairment, 10-20 indicating moderate impairment, and 21-26 indicating mild impairment.
Modified Barium Swallow Impairment Profile | day 1 and day 14
  Modified Barium Swallow Impairment Profile is a scale used to assess swallowing dysfunction.The scale assesses various aspects of swallowing by observing the patient's swallowing actions during a videofluoroscopic swallow study, including oral phase, pharyngeal transit, swallow delay, and upper esophageal sphincter opening. Scores on the Modified Barium Swallow Impairment Profile range from 0 to 55, with higher scores indicating more severe impairment.
Functional Oral Intake Scale | day 1 and day 14
  During Dysphagia-Functional Oral Intake Scale assessment, evaluators engage in communication with the patient, conduct observations, and make records to assess the patient's oral intake ability. The Functional Oral Intake Scale assessment form includes seven levels of scoring, ranging from level 1 to level 7, indicating a progressive improvement in the patient's oral intake ability. In general, the result below level 6 indicates unsafe for oral intake while level 6 and above indicates that eating via mouth can be safely conducted.

CONTACTS AND LOCATIONS:
Overall Officials: Nieto Luis, Master, Principal Investigator — Site Coordinator of United Medical Group
Locations (3):
- China (3):
  - Affiated Hos. Campus of zdy, Zhongguo
  - River south medical affili. Campus of zdy, Zhongguo
  - The 4th affili. (Huij) Campus of zdy, Zhongguo

IPD SHARING:
Plan to Share IPD: No